CLINICAL TRIAL: NCT03380806
Title: A Randomized Phase II Trial Investigating Stereotactic Body RadioTherapy (SBRT) for Prostate Boost Irradiation in the Treatment of High Risk Prostate Cancer (PrCa)
Brief Title: Prostate Boost Irradiation With Stereotactic Body RT (SBRT)
Acronym: PBS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juravinski Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Naghmeh Isfahanian, Term Professional staff, Juravinski Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4178
Record Dates: First submitted 2017-12-13; First posted 2017-12-21 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
Keywords: stereotactic body radiotherapy (SBRT); conventional radiotherapy (CRT); High risk prostate cancer; quality of life (QoL); The Expanded Prostate cancer Index Composite (EPIC-26); International Prostate Symptom Score (IPSS)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; luprolide acetate gel depot; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Conventional Radiotherapy (CRT) Prostate Boost Pelvic Radiation LHRH agonist
  Interventions: Drug: LHRH agonist; Radiation: Pelvic Radiation; Radiation: Conventional Radiotherapy (CRT) Prostate Boost
- Arm 2 (Experimental): Stereotactic Body Radiotherapy (SBRT) Prostate Boost Pelvic Radiation LHRH agonist
  Interventions: Drug: LHRH agonist; Radiation: Pelvic Radiation; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: LHRH agonist — Standard LHRH agonist for 3 years
  Other Names: Eligard
Radiation: Pelvic Radiation — Pelvic Radiation
Radiation: Stereotactic Body Radiotherapy (SBRT) — SBRT: 19.5 - 21 Gy in three fractions (1 treatment per week - over 22days)
  Arms: Arm 2
Radiation: Conventional Radiotherapy (CRT) Prostate Boost — CRT: 33 - 35 Gy in 16 fractions (5 days per week - over 22 days)
  Arms: Arm 1

SUMMARY:
A randomized controlled open-label trial in patients with high risk prostate cancer. Eligible and consenting patients will be randomly allocated to receive stereotactic body radiotherapy (SBRT) boost to prostate or conventional radiotherapy boost to prostate in 1:1 ratio. Prostate radiotherapy boost will be administered after standard pelvic radiotherapy. Subjects will be followed for 24 months post radiation treatment for Quality of Life assessment and toxicity.

DETAILED DESCRIPTION:
In this study we investigate stereotactic body radiotherapy (SBRT) as a boost radiotherapy treatment, following pelvic radiotherapy, in patients with high risk prostate cancer (PrCa) treated with Androgen Deprivation Therapy (ADT). One hundred patients with localized high risk PrCa will receive ADT for a total of 3 years. Three months after initiation of ADT all patients will receive pelvic (lymph node and prostate) treatment of 45Gy in 25 fractions (5 days per week). Then patients will be randomized to receive either The conventional radiotherapy (CRT) of 33 - 35 Gy in 16 fractions (5 days per week - over 22 days) (comparator arm) or SBRT boost treatment of 19.5 - 21 Gy in three fractions (1 treatment per week - over 22days) (experimental arm). SBRT boost treatment will be delivered with either cyberknife or VMAT technique.

ELIGIBILITY:
Inclusion Criteria:

* Histological and or clinical diagnosis of high risk adenocarcinoma of the prostate within six months of entry (stage T3 or higher and/or Gleason score 8 or higher and/or initial PSA level above 20;)
* No radiographic evidence of metastatic disease to the abdomen, lymph nodes, bone or other distant organs; determined by standard staging investigations (bone scan and CT-scan of the abdomen and pelvis) or incidental findings (localized N0, M0 disease)
* Patient is able to complete the quality of life questionnaires in English.
* Informed consent obtained

Exclusion Criteria:

* • Histological diagnosis of carcinoma of the prostate more than six months prior to potential registration date;
* Previous treatment for carcinoma of the prostate (other than biopsy or TURP), including bilateral orchiectomy;
* Patients previously on more than twelve weeks of hormone therapy for their PrCa;
* Past history of other malignancies except: adequately treated non-melanoma skin cancer or other solid tumours curatively treated with no evidence of disease for more than 3 years;
* Contraindications to placement of gold seeds for daily prostate localization;
* Previous pelvic RT and/or significant pelvic surgery;
* Severe diverticular or inflammatory bowel disease (as determined by the treated radiation oncologist)
* Previous hip replacement
* PSA over 50
* IPSS 20 or higher
* TRUS-based prostate
* volume of > 80 cc

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Short Term Quality of Life (QoL) | up to 6 months post radiation
  To compare early QoL (up to 6 months post RT) in patients with high risk adenocarcinoma of the prostate treated with ADT and RT in the form of pelvic nodal irradiation and prostate boost with standard fractionation, or pelvic nodal irradiation and prostate boost with SBRT using Cyberknife or VMAT. QoL, defined as bowel and bladder function and bother after PrCa treatment, will be measured prior to and at regular intervals after completion of radiotherapy using the established Prostate QoL (The Expanded Prostate cancer Index Composite (EPIC-26 instrument)). Higher EPIC score represent a better outcome

SECONDARY OUTCOMES:
Long Term Quality of Life (QoL) | 24 months
  long term QoL QoL, defined as bowel and bladder function and bother after PrCa treatment, will be measured prior to and at regular intervals up to 24 months month after completion of radiotherapy using the established Prostate QoL (The Expanded Prostate cancer Index Composite (EPIC-26 instrument)). Higher EPIC score represent a better outcome
Urinary function assessment | 24 months
  short and long term quality of urinary function (The International Prostate Symptom Score (IPSS)).
  Total IPSS is between 1-35 / lower score shows better function.
Late Toxicity | 12-24 months
  Grade 2-4 treatment related late (12-24 months), bladder and bowel related toxicity evaluated by the Expanded Common Toxicity Criteria of the National Cancer Institute of Canada (NCI)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Walker Family Cancer Centre ,Niagara Health - St. Catharines Site, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gouveia A, Mesci A, Isfahanian N, Dayes I, Quan K, Goldberg M, Schnarr KL, Lukka H, Cuthbert D, Hallock A, Douvi G, Wright J, Swaminath A, Chow T, Diamond K, Hajdok G, Maharaj L, Ewusie J, Tsakiridis T. Primary Analysis of (NCT03380806) a Phase II Randomized Trial of Stereotactic Body Radiotherapy Boost Versus Conventional Fractionation External Beam Radiotherapy Boost in Unfavorable-Intermediate and High-Risk Prostate Cancer. Prostate. 2025 Jul;85(10):977-985. doi: 10.1002/pros.24905. Epub 2025 Apr 27. PMID 40287937